CLINICAL TRIAL: NCT02085031
Title: Randomized Controlled Trial on Surgical Safety of Intracorporeal Versus Extracorporeal Roux-en-Y Esophagojejunostomy During Laparoscopic Total Gastrectomy for Gastric Cancer
Brief Title: Intracorporeal Versus Extracorporeal Roux-en-Y Esophagojejunostomy During Laparoscopic Total Gastrectomy for Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Li, M.D., Ph.D., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFGS-OrVil-01
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Stomach Neoplasms; Minimally Invasive Surgery; Anastomosis
Keywords: Roux-en-Y Anastomosis; laparoscopic surgery; minilaparotomy; stomach neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracorporeal Roux-en-Y esophagojejunostomy (Experimental): During totally laparoscopic total gastrectomy, Roux-en-Y esophagojejunostomy intracorporeally using a transorally inserted anvil (OrVil™) will be performed for the patients assigned to this arm.
  Interventions: Procedure: Intracorporeal Roux-en-Y esophagojejunostomy
- Extracorporeal Roux-en-Y esophagojejunostomy (Active Comparator): During laparoscopic total gastrectomy, Roux-en-Y esophagojejunostomy extracorporeally using a transabdominally inserted anvil will be performed for the patients assigned to this arm.
  Interventions: Procedure: Extracorporeal Roux-en-Y esophagojejunostomy

INTERVENTIONS:
Procedure: Intracorporeal Roux-en-Y esophagojejunostomy — During totally laparoscopic total gastrectomy, Roux-en-Y esophagojejunostomy intracorporeally using a transorally inserted anvil (OrVil™) will be performed.
  Arms: Intracorporeal Roux-en-Y esophagojejunostomy
Procedure: Extracorporeal Roux-en-Y esophagojejunostomy — During laparoscopic total gastrectomy, Roux-en-Y esophagojejunostomy extracorporeally using a transabdominally inserted anvil will be performed.
  Arms: Extracorporeal Roux-en-Y esophagojejunostomy

SUMMARY:
* To date, Roux-en-Y esophagojejunostomy transabdominal extracorporeally by circular stapler was the most common used method during laparoscopy-assisted total gastrectomy for gastric cancer, even though it was not totally laparoscopic surgery in which intracorporeal anastomosis should be performed.
* To gain potential clinical benefits from a smaller length of minilaparotomy and an easier anastomosis technique than extracorporeal anastomosis, intracorporeal Roux-en-Y anastomosis using a transorally inserted anvil (OrVil™) during totally laparoscopic total gastrectomy was adopted by experienced surgeons recently.
* However, the safety of intracorporeal Roux-en-Y esophagojejunostomy using a transorally inserted anvil (OrVil™) has not yet been evaluated. Thus, the study comparing the safety of intracorporeal versus extracorporeal Roux-en-Y esophagojejunostomy by circular stapler based on a well designed randomized controlled trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma confirmed pathologically by endoscopic biopsy
* Tumor located at middle or upper third of stomach while laparoscopic total gastrectomy is the planning surgery
* Tumor invasion is less than 3cm above the esophagogastric junction
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* Conversion to open surgery before reconstruction

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Anastomosis-related early complication rate | 30 days
  Anastomotic leakage, intraluminal bleeding, or stenosis were considered as anastomosis-related early complication.

SECONDARY OUTCOMES:
Reconstruction time | During operation
  Experimental group (Intracorporeal group): time from the esophagus was transected to reconstruction was completed.
  Active Comparator (Extracorporeal group): time from the minilaparotomy was made to reconstruction was completed.
Morbidity and mortality rates | 30 days
  The early postoperative complication was defined as the event observed within 30 days after surgery.
Postoperative recovery course | 2 weeks
  Time to first ambulation, flatus, liquid diet, soft diet, and postoperative hospital stay were used to assess the postoperative recovery course.
Postoperative quality of life | 6 months
  EORTC questionaire (STO-22 and C30) were used to access the postoperative quality of life at 0,1,3,6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University, China
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Marangoni G, Villa F, Shamil E, Botha AJ. OrVil-assisted anastomosis in laparoscopic upper gastrointestinal surgery: friend of the laparoscopic surgeon. Surg Endosc. 2012 Mar;26(3):811-7. doi: 10.1007/s00464-011-1957-x. Epub 2011 Oct 13. PMID 21993942
- [Background] Jeong O, Park YK. Intracorporeal circular stapling esophagojejunostomy using the transorally inserted anvil (OrVil) after laparoscopic total gastrectomy. Surg Endosc. 2009 Nov;23(11):2624-30. doi: 10.1007/s00464-009-0461-z. Epub 2009 Apr 3. PMID 19343421
- [Background] Kunisaki C, Makino H, Oshima T, Fujii S, Kimura J, Takagawa R, Kosaka T, Akiyama H, Morita S, Endo I. Application of the transorally inserted anvil (OrVil) after laparoscopy-assisted total gastrectomy. Surg Endosc. 2011 Apr;25(4):1300-5. doi: 10.1007/s00464-010-1367-5. Epub 2010 Oct 17. PMID 20953884
- [Background] Jeong O, Jung MR, Kim GY, Kim HS, Ryu SY, Park YK. Comparison of short-term surgical outcomes between laparoscopic and open total gastrectomy for gastric carcinoma: case-control study using propensity score matching method. J Am Coll Surg. 2013 Feb;216(2):184-91. doi: 10.1016/j.jamcollsurg.2012.10.014. Epub 2012 Dec 2. PMID 23211117
- See also: Southern Medical University, China — http://www.fimmu.com/index_com.html
- See also: Nanfang Hospital, China — http://www.nfyy.com
- See also: Chinese Anti-Cancer Association — http://www.caca.org.cn